CLINICAL TRIAL: NCT05680818
Title: CALIBRATE: A Phase 3, Randomized, Open-Label Study Evaluating the Efficacy and Safety of Encaleret Compared to Standard of Care in Participants With Autosomal Dominant Hypocalcemia Type 1 (ADH1)
Brief Title: Efficacy and Safety of Encaleret Compared to Standard of Care in Participants With ADH1
Acronym: CALIBRATE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Calcilytix Therapeutics, Inc., a BridgeBio company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLTX-305-302
Record Dates: First submitted 2022-12-12; First posted 2023-01-11 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Autosomal Dominant Hypocalcemia (ADH)
Keywords: Autosomal Dominant Hypocalcemia Type 1 (ADH1); Hypocalcemia; Musculoskeletal Diseases; Muscular Diseases; Musculoskeletal Abnormalities; Calcium Metabolism Disorders; Metabolic Diseases; Hypoparathyroidism; Hypocalcemic Seizures; Hypercalciuria; Nephrocalcinosis; Nephrolithiasis; Calcium Sensing Receptor; Encaleret; Hypopara
MeSH Terms: conditions — Hypercalciuric Hypocalcemia, Familial; Hypocalcemia; Musculoskeletal Diseases; Muscular Diseases; Musculoskeletal Abnormalities; Calcium Metabolism Disorders; Metabolic Diseases; Hypoparathyroidism; Hypercalciuria; Nephrocalcinosis; Nephrolithiasis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Encaleret (Experimental): Participants will receive encaleret at a dose as needed based on calcium levels.
  Interventions: Drug: Encaleret
- Standard of Care (SoC) (Other): Participants will continue receiving calcium supplements and/or active Vitamin D (calcitriol, alfacalcidol, falecalcitriol, etc.)
  Interventions: Dietary Supplement: Standard of Care

INTERVENTIONS:
Drug: Encaleret — Administered as film-coated tablet for oral use
  Other Names: CLTX-305; Encaleret Sulfate
  Arms: Encaleret
Dietary Supplement: Standard of Care — Calcium supplements and/or active Vitamin D (calcitriol, alfacalcidol, falecalcitriol, etc.)
  Arms: Standard of Care (SoC)

SUMMARY:
The primary purpose of the study is to understand the effectiveness, safety, and tolerability of encaleret when compared to standard of care (SoC) treatment in participants with Autosomal Dominant Hypocalcemia Type 1 (ADH1).

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants must have a documented pathogenic or likely pathogenic activating variant, or variant of uncertain significance, of the calcium sensing receptor (CASR) gene associated with biochemical findings of hypoparathyroidism.
2. Participants must have a documented history of symptoms or signs of ADH1.
3. Participants 16 to <18 years old must have closed growth plates on hand radiograph.
4. Participants treated with thiazide diuretics must discontinue thiazides for at least 14 days prior to SoC Optimization Visit 1 through Week 24 (Period 3). When the thiazide is being used as an antihypertensive, alternative therapy will be prescribed by the Investigator as needed.
5. Participants treated with phosphate binders (other than calcium salts) must discontinue the phosphate binders at least one day prior to the SoC Optimization Visit 1.
6. Participants treated with magnesium or potassium supplements must be willing to discontinue such treatment prior to the first dose of encaleret.
7. Participants treated with potassium-sparing diuretics must be willing to discontinue such treatment prior to the first dose of encaleret.
8. Participants must meet SoC Optimization criteria as defined in the protocol.

Key Exclusion Criteria:

1. History of hypocalcemic seizure within the past 3 months preceding Screening.
2. History of thyroid or parathyroid surgery.
3. History of renal transplantation.
4. Pregnant or nursing (lactating) women, where pregnancy is confirmed by a positive beta-human chorionic gonadotropin (β-hCG) laboratory test.
5. History of treatment with parathyroid hormone (PTH) 1-84 or 1-34 within the 2 months preceding Screening and requiring SoC doses exceeding >1.2× their pre-PTH treatment total daily doses or bone turnover markers, Collagen cross-linked C-telopeptide (CTx )and Procollagen type 1 N-propeptide (P1NP), > upper limit of normal for sex, age (men only) and menopausal status (women only).
6. Blood 25-OH Vitamin D level <25 nanograms (ng)/milliliter (mL).
7. Estimated glomerular filtration rate (eGFR) <30 mL/minute/1.73 m^2 using chronic kidney disease-EPI creatinine equation refit without the race variable (chronic kidney disease-EPI creatinine equation refit without the race variable [CKD-EPIcr_R]) (for participants <18 years old the Bedside Schwartz equation should be used).
8. Participants with positive Hepatitis B surface antigen (HBsAg), Hepatitis A immunoglobulin M (IgM), or human immunodeficiency virus (HIV) viral serology test at the Screening Visit. Participants who are in complete remission from Hepatitis C virus (HCV) as evidenced by sensitive assay ≥12 weeks after completion of HCV therapy may participate in the study.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Number of Responders who Achieve Both Albumin-Corrected Blood Calcium (cCa) and 24-hour Urinary Calcium (UCa) Within the Target Range | Up to Week 24
  * cCa within 8.3-10.7 mg/dL (2.08-2.68 millimoles per liter [mmol/L])
  * 24-hr UCa within the reference range (< 300 mg/day for men [7.5 mmol/day], < 250 mg/day for women [6.25 mmol/day])

SECONDARY OUTCOMES:
Number of Participants With Intact Parathyroid Hormone (iPTH) Within or Greater than the Reference Range | Up to Week 24
Number of Participants who Achieve Blood Magnesium Within the Reference Range | Up to Week 24
Number of Participants who Achieve Blood Phosphate Within the Reference Range | Up to Week 24
Change From Baseline in Blood 1,25-(OH)2 Vitamin D | Baseline to Week 24
Change From Baseline in cCa | Baseline to Week 24
Change From Baseline in 24-hour UCa | Baseline to Week 24
Change From Baseline in iPTH | Baseline to Week 24
Change From Baseline in Blood Phosphate and Blood Magnesium | Baseline to Week 24
Change From Baseline in Urine Magnesium, Phosphate, Sodium, and Citrate Handling | Baseline to Week 24
Change From Baseline in QT Interval Corrected for Changes in the Heart Rate With Fridericia Formula (QTcF) as Assessed by Electrocardiogram (ECG) | Baseline to Week 24
Change from Baseline in 36-Item Short Form Health Survey (SF-36) Physical Component Score and Mental Component Score and Each of the Sub-Domains | Baseline to Week 24
Number of Participants in the Encaleret Arm Receiving Calcium and/or Vitamin D Supplements | Up to Week 24
Steady State Encaleret Trough Concentration (Ctrough) | Up to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Calcilytix Medical Director, Study Director — Calcilytix Therapeutics, Inc., a BridgeBio company
Locations (25):
- United States (11):
  - UCSF Benioff Children's Hospital, Oakland, Oakland, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - NIH, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Columbia University Irving Medical Center, New York, New York
  - Physicians East, Greenville, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Houston Methodist Hospital, Houston, Texas
- Australia (2):
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
- Bone Research & Education Centre, Oakville, Ontario, Canada
- Vseobecna fakultni nemocnice v Praze, New Town, Czechia
- Aarhus University Hospital, Aarhus, Denmark
- France (2):
  - CHU Bicetre, Le Kremlin-Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Edouard Herriot - HCL, Lyon
- Italy (3):
  - IRCCS Ospedale San Raffaele, Milan
  - University Hospital of Pisa, Pisa
  - Fondazione Policlinico Universitario Campus Bio-Medico, Roma
- The University of Tokyo Hospital, Tokyo, Japan
- Eramus MC, Rotterdam, Netherlands
- United Kingdom (2):
  - Freeman Hospital, Newcastle upon Tyne
  - Norfolk and Norwich University Hospital, Norwich

IPD SHARING:
Plan to Share IPD: No